CLINICAL TRIAL: NCT07391527
Title: Early Detection and Prevention of Health Complications in Premature Infants - Early Detection of Developmental Abnormalities of Preterm Infants at 5 Years of Age
Brief Title: Early Detection of Developmental Abnormalities of Preterm Infants at 5 Years of Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: České Budějovice Hospital (Other); General University Hospital, Prague (Other); Hospital Havlickuv Brod (Unknown); County Hospital Liberec, Liberec (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UZIS 2025/3
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: 5 Year Old Children Born Prematurely
Keywords: follow up of premature infants; early detection; developmental abnormality; Czech Republic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5 year old children born prematurely (Other)
  Interventions: Other: Pediatric check-up

INTERVENTIONS:
Other: Pediatric check-up — Eligible children are invited to undergo a comprehensive pediatric evaluation, including vision screening (Plusoptix) and speech and language tests (TEPO - sentence comprehension, TEPRO - vocabulary production). Subsequently, children are referred for psychological (IDS-P), motor (MABC-2), and pulmonary (spirometry) assessments. If any deviations are identified, the child is referred to appropriate specialists (e.g., rehabilitation physician, speech therapist, psychiatrist, ophthalmologist).

SUMMARY:
The project is a national, prospective, multicenter, interventional pilot project focused on the follow up of 5 year old children that were born prematurely.

The primary aim of the project is to prepare, test, and develop a proposal for a national methodology for the care of children born prematurely. This will minimize the negative impacts on the overall development of the child and the family of the prematurely born children.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, interventional pilot project focused on the follow up of 5 year old children that were born prematurely.

The main goal of the project is establishing a methodology for the long-term monitoring of premature infants (in the area of developmental anomalies) and their evaluation at the age of 5 years.

The main objective of this activity is to validate this screening process, which will benefit 210 patients in 2 perinatal and 2 intermediate centers. The child will undergo a comprehensive pediatric examination, including basic vision, speech, and psychomotoric assessments (MABC-2 and IDS-P). If any concerns are identified, the child will be referred to an appropriate specialist. The timeliness of this check-up has significant positive impact on both the patient and their family.

The project is supported by the European Social Fund (Operational Program Employment plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0002020.

The study has been reviewed and approved by multiple local ethical committees. The listed IRB represents the lead national ethical committee overseeing the trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent for participation in the project and consent for the processing of personal data.
* Children born before 37 weeks of gestation, aged 5 years, growing up in a Czech-speaking environment.
* To ensure valid linkage of all data sources, the children must have been born to parents with Czech citizenship.

Exclusion Criteria:

* Unsigned consent for participation in the project and consent for the processing of personal data.
* Severe psychomotor retardation .
* Severe congenital malformations.

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of premature infants with identified pathology at 5 years (overall, by detected pathology) | During study participation (up to 3 days)
Proportion of premature infants referred to a specialized center (overall, by detected pathology) | During study participation (up to 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Marková, M.D., Study Director — General Hospital University in Prague; Richard Plavka, prof., Study Director — General Hospital University in Prague
Locations (4):
- Czechia (4):
  - České Budějovice Hospital, České Budějovice, Czech Republic
  - Hospital Havlíčkův Brod, Havlíčkův Brod, Czech Republic
  - County Hospital Liberec, Liberec, Czech Republic
  - General University Hospital, Prague, Czech Republic

IPD SHARING:
Plan to Share IPD: No